CLINICAL TRIAL: NCT04582097
Title: Impact of Angiotensin-converting Enzyme Inhibitor on Pediatric Hemodialysis Patients
Brief Title: Ramipril in Pediatric Patients on Hemodialysis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Areej Mohamed Ateya, Assisstant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHCL 65
Record Dates: First submitted 2020-10-03; First posted 2020-10-09 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Hemodialysis
Keywords: angiotensin-convertting enzyme inhibitor; ramipril
MeSH Terms: interventions — Ramipril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ramipril (Experimental): Ramipril, 2.5 mg daily, administered orally for 16 weeks
  Interventions: Drug: Ramipril
- Placebo (Placebo Comparator): Placebo, matched for the interventional drug, administered orally, daily for 16 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ramipril — angiotensin-converting enzyme inhibitor
  Other Names: Tritace
  Arms: Ramipril
Drug: placebo — same odor, color and size as the drug but without the active ingredient
  Arms: Placebo

SUMMARY:
The aim of the study is to evaluate the effect of Ramipril in pediatric patients on regular hemodilaysis

DETAILED DESCRIPTION:
Evaluate the effect of Ramipril on blood pressure, heart rate, Endothelial dysfunction and inflammatory markers in pediatric patients on regular hemodilaysis and the correlation of response with ACE I/D polymorphisms.

ELIGIBILITY:
Inclusion Criteria:

* Patients < 16 years old
* Patients who have been on regular HD for 6 months or longer
* Hypertension at enrollment

Exclusion Criteria:

* History of active connective tissue disease
* Acute infection within 1 month prior to the study
* Advanced liver disease
* Gastrointestinal dysfunction requiring parental nutrition or active malignancy
* Use of medications such as immunosuppressive drugs within 1 month prior to the study
* Use of anti-inflammatory medications
* Use of vitamin E at a dose higher than 60 IU per day or vitamin C higher than 500 mg per day
* History of myocardial infarction or cerebrovascular event within 3 months prior to the study
* History of ACE inhibitor-associated angioedema
* Inability to discontinue ACE inhibitors or ARBs

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
concentration of Asymmetric dimethylarginine (ADMA) | 16 weeks
  marker of endothelial dysfunction
concentration of high-sensitivity C-reactive protein (Hs-CRP ) | 16 weeks
  marker of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Ain Sh University, Principal Investigator — university
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ateya AM, El Hakim I, Shahin SM, El Borolossy R, Kreutz R, Sabri NA. Effects of Ramipril on Biomarkers of Endothelial Dysfunction and Inflammation in Hypertensive Children on Maintenance Hemodialysis: the SEARCH Randomized Placebo-Controlled Trial. Hypertension. 2022 Aug;79(8):1856-1865. doi: 10.1161/HYPERTENSIONAHA.122.19312. Epub 2022 Jun 10. PMID 35686561